CLINICAL TRIAL: NCT02274025
Title: Collection of Lung Malignant Tissue for the Validation of a Novel Technology to Identify Oncogenic Mutations and Personalized Medicine
Brief Title: NovellusDx Functional Profiling of Oncogenic Mutations in Lung Cancer Patients
Status: Completed | Type: Observational
Sponsor: Fore Biotherapeutics (Industry)
Collaborators: Rabin Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: TISS001
Record Dates: First submitted 2014-10-14; First posted 2014-10-24 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2015-10

CONDITIONS: Lung Cancer
Keywords: Patient diagnosed with lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Biopsy material of patient or pleural fluids.
Oversight: Data Monitoring Committee: No

SUMMARY:
NovellusDx technology identifies tumor-specific driver mutations, but unlike sequencing-based tests, NovellusDx has a functional assay that detects dis-regulated translocation of mutated signaling proteins to the nucleus. This allows NovellusDx to identify functionally-impactful driver mutations regardless of whether the mutation has previously been described or linked to a tumor type.

ELIGIBILITY:
Inclusion Criteria:

* Patients that are suspected to have lung cancer and are eligible for biopsy, surgical intervention or pleural fluid suction

Exclusion Criteria:

* Patients without lung cancer

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that are suspected to have lung cancer and are eligible for biopsy, surgical intervention or pleural fluid suction.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Correct identification of tumor mutant genes | up to 12 months
  Correct identification of patient oncogenic mutation in over 85% of the cases. this will be achieved by comparing sequencing results of the patient tumors to the results achieved using the NovellusDx diagnostic platform.

CONTACTS AND LOCATIONS:
Overall Officials: Mordechai Kremer, Prof, Principal Investigator — Rabin Medical Center, Beilinson
Locations (1):
- Rabin Medical Center, Beilinson, Petah Tikva, Israel